CLINICAL TRIAL: NCT01647256
Title: Comparison of Nikkomycin Z Bioavailability After Single Dose Administration Under Fed (High Fat Meal) Compared to Fasting Conditions
Brief Title: Comparison of Nikkomycin Z Bioavailability Under Fed and Fasting Conditions
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient # subjects available for 2nd group; evaluating alternate study site
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VFCE-2011-004
Record Dates: First submitted 2012-07-16; First posted 2012-07-23 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: Bioavailability; Fed; Fasting
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency; Fasting | interventions — nikkomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nikkomycin Z fed - fasting (Experimental): Period 1:
  * Day 1: Nikkomycin Z 500 mg with high fat breakfast
  Period 2:
  * Day 1: Nikkomycin Z 500 mg under fasted conditions
  Interventions: Drug: Nikkomycin Z
- Nikkomycin Z fasting - fed (Experimental): Period 1:
  * Day 1: Nikkomycin Z 500 mg under fasted conditions
  Period 2:
  * Day 1: Nikkomycin Z 500 mg with high fat breakfast
  Interventions: Drug: Nikkomycin Z

INTERVENTIONS:
Drug: Nikkomycin Z — Capsule, 500 mg, single-dose

SUMMARY:
The primary purpose of this study is to evaluate if eating a high fat meal versus not eating any food affects how the study drug (Nikkomycin Z) is absorbed into the body. The second purpose is to gain further information about the safety of Nikkomycin Z in healthy adults.

DETAILED DESCRIPTION:
To compare the single-dose bioavailability of Nikkomycin Z 500 mg (two 250 mg capsules) under fed and fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age and not over 40 years of age
* Be male, or female (non childbearing potential or using adequate contraception)
* Have a body mass index between 18 and 29 kg/m2
* Able to understand the study and give written informed consent
* Be determined healthy based on a medical and laboratory evaluation

Exclusion Criteria:

* Patients under the age of 18 years or over 40 years of age
* Current smoker or history of smoking within 3 months of participation
* Inability to comprehend study and provide written informed consent
* Inability to comply with the study requirements
* History of or current evidence of major organ disease
* Renal disease - serum creatinine > 1.5 mg/dL, significant hematuria or proteinuria, known structural abnormality or chronic kidney disease
* Hepatic disease - active viral hepatitis, history of hepatitis B or hepatitis C, bilirubin > 2.0, ALT or AST above normal upper limit for laboratory, alcoholic liver disease, other chronic liver disease
* CNS disease or cognitive dysfunction - any past history of epilepsy, CNS infections, stroke, CNS bleed, severe headaches, major psychiatric illness, or current mental status changes
* Lung disease - history of severe asthma, COPD, pulmonary tuberculosis, or other major lung disease
* Cardiac disease - history or current evidence of ischemic coronary artery disease, myocardial infarction, heart failure, or significant arrhythmia
* Gastrointestinal disease - presence of inflammatory bowel disease, difficulty swallowing, or any gastrointestinal probably that would limit taking oral medications or that may compromise absorption of oral medications
* Cancer - History of hematologic malignancy or solid tumor excluding basal cell carcinoma limited to the skin within the past 5 years
* History of autoimmune or inflammatory disease such as rheumatoid arthritis and lupus
* Immunocompromised state - solid organ transplant, cancer chemotherapy, stem cell transplant with graft versus host disease, immunosuppressive therapy, or HIV infection
* Recent weight loss of greater than 10%
* Any other history or evidence of disease that in the opinion of the physician would increase the risk for the subject for clinical trial participation
* Regular use of prescription medications, over-the-counter medications, or dietary/herbal supplements within 14 days of day 1. Occasional use of acetaminophen or over-the-counter NSAID within the 14 day window may be allowed at the P.I. discretion
* Subjects who received another investigational drug within 30 days of enrollment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Rate and extent of Nikkomycin Z absorption under fed and fasting conditions | 24 hours

SECONDARY OUTCOMES:
Extent of Nikkomycin Z urinary excretion | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn R Matthias, PharmD, Principal Investigator — University of Arizona; David E Nix, PharmD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona - Clinical and Translational Science Research Center, Tucson, Arizona, United States